CLINICAL TRIAL: NCT00392951
Title: Sirolimus for Patients With Chronic and/or Refractory Autoimmune Cytopenias: A Pilot Series
Brief Title: Sirolimus for Autoimmune Disease of Blood Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-7-4873
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Autoimmune Pancytopenia; Autoimmune Lymphoproliferative Syndrome (ALPS); Evans Syndrome; Idiopathic Thrombocytopenic Purpura; Anemia, Hemolytic, Autoimmune; Autoimmune Neutropenia; Lupus Erythematosus, Systemic; Inflammatory Bowel Disease; Rheumatoid Arthritis
Keywords: ALPS; Autoimmune; Cytopenias; Treatment; Sirolimus; Rapamycin; Lymph Nodes; Spleen; Hemolytic Anemia; Immune Thrombocytopenia; Neutropenia; ITP; Lupus
MeSH Terms: conditions — Autoimmune Lymphoproliferative Syndrome; Evans Syndrome; Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune; Lupus Erythematosus, Systemic; Inflammatory Bowel Diseases; Arthritis, Rheumatoid; Cytopenia; Anemia, Hemolytic; Neutropenia | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus treatment (Experimental): Sirolimus treatment
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — Tablet or liquid; taken once or twice daily; dosage is based on establishing a serum trough of 5-15 ng/ml by high-performance liquid chromatography (initial loading dose of 3 mg/m2 then 2.5 mg/m2 with adjustment based on serum trough)
  Other Names: rapamycin; rapamune

SUMMARY:
Treatment for patients with autoimmune destruction of blood cells is poor. The part of the body that fights infections is called the immune system and white blood cells (WBCs) are part of the immune system. Normally, a person's body creates WBCs to fight infections and eliminates WBCs which have stopped helping the body function. Patients with autoimmune destruction of blood cells have difficulty eliminating old WBCs. The abnormal WBCs build up and can damage other healthy cells, which can lead to anemia, fatigue, jaundice, internal bleeding, infection, and cancer. Few effective medications exist for treatment for patients with autoimmune cytopenias and those commonly used are fraught with side effects. Nevertheless, as scientific understanding of autoimmune diseases has improved, more directed and less toxic therapies are becoming available. A number of groups have been studying the efficacy of a medication called sirolimus in patients with autoimmune diseases. This medicine has been FDA-approved for over 20 years. Sirolimus is a medicine used in children with other diseases. Sirolimus works, in part, by eliminating old and abnormal WBCs. Our group and others have shown that sirolimus is effective in mice with autoimmunity and in children with a rare condition called Autoimmune Lymphoproliferative Syndrome (ALPS). We believe sirolimus will help children with autoimmune cytopenias. We believe it will improve their symptoms and make them less sick. We propose to study sirolimus in children with chronic and/or refractory autoimmune cytopenias.

DETAILED DESCRIPTION:
Patients with autoimmune destruction of hematopoietic cells frequently have severe and debilitating disease requiring aggressive and frequent medical management. These patients are often treated with non-specific immunosuppressive medications with limited efficacy and untoward side-effect profiles. We have been investigating the use of an immunosuppressive and anti-cancer agent, sirolimus in patients with an autoimmune cytopenias syndrome: Autoimmune Lymphoproliferative Syndrome (ALPS). ALPS is a primary immune deficiency caused by mutations in the Fas apoptotic pathway, leading to abnormal lymphocyte survival. Clinical manifestations in patients with ALPS typically include autoimmune cytopenias, lymphadenopathy, hepatosplenomegaly, and a propensity to develop secondary malignancies. Thus, far we have found excellent results albeit the total number of patients treated is small.

Sirolimus is a signal transduction inhibitor with a tolerable side effect profile. Sirolimus has two properties making it an attractive agent to treat patients with autoimmune cytopenias syndromes, including ALPS. First, sirolimus induces apoptosis in normal and abnormal white blood cells, the cell type dysregulated in patients with autoimmune disease. In addition, sirolimus increases a T cell subset called Regulatory T cells (Tregs). Tregs are a cell population designed to suppress the immune system and control autoimmunity. These combined properties make sirolimus unique as compared with other immunosuppressive agents. Ample preclinical and clinical data exists demonstrating sirolimus in effective in patients with autoimmunity. Accordingly, we hypothesize sirolimus is a safe and efficacious medication for patients with autoimmune destruction of blood cells..

We plan to confirm our hypotheses by performing a pilot series in children with autoimmune cytopenias who are either refractory to standard therapy or have significant toxicity from standard treatments. Our primary aim is to define the toxicities of administration of oral sirolimus in children with autoimmune cytopenias. Our secondary aims are to evaluate the efficacy of sirolimus in children with autoimmune cytopenias, to determine the trough levels of sirolimus when used in these patients, and to evaluate the effects of sirolimus on intracellular targets of mammalian target of rapamycin (mTOR). We intend to enroll 50 children with autoimmune cytopenias and treat for a 6 month period, however, if we find sirolimus is effective, we anticipate these children will continue to take sirolimus for a longer period of time. We anticipate the results of this work will establish sirolimus is an effective and well tolerated medication and will lead directly to a larger national phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 months and < 30 years at the time of study entry
* Diagnosis of autoimmune cytopenias requiring treatment with medications
* At least one of the following: Autoimmune Neutropenia, Autoimmune Hemolytic Anemia, and/or Autoimmune Thrombocytopenia
* Must be proven autoimmune by either a documented autoantibody (positive direct anti globulin test, positive anti-neutrophil, and/or anti-platelet antibody) and/or a documented clinical response to immunosuppression
* Autoimmune Cytopenias can be idiopathic (Idiopathic Thrombocytopenic Purpura (ITP), Autoimmune Hemolytic Anemia (AIHA), Autoimmune Neutropenia (AIN), or Evans syndrome) or secondary to one of following conditions: Lupus, Rheumatoid Arthritis (RA), ALPS (Autoimmune Lymphoproliferative Syndrome), or Inflammatory bowel disease (IBD)
* Patients must have chronic disease diagnosed by either a documented cytopenia syndrome (Lupus, ALPS, RA, or IBD), or by having Evans syndrome defined as idiopathic destruction of multiple blood cell types, and/or by having disease >6 months
* Patients must be refractory to or unable to tolerate standard front-line therapies for autoimmune cytopenias (corticosteroids and/or IVIG)
* Patients may be taking second-line agents for autoimmune cytopenias (mycophenolate mofetil, cyclosporine, tacrolimus, mercaptopurine, and/or methotrexate) at time of study entry; however, attempts should be made to wean these agents. Patients may not stay on a combination of sirolimus and a calcineurin inhibitor for greater than 4 weeks
* Informed consent/assent must be obtained prior to initiating treatment
* Patient must be able to consume oral medication in the form of tablets or solution

Exclusion Criteria:

* Pregnancy or breast feeding
* Uncontrolled infection
* Known allergy to Sirolimus or its components
* Patients with a documented malignancy on therapy or not in remission
* Patients who do not meet organ function requirements listed in protocol
* Patients with a documented history of severe combined immunodeficiency or human immunodeficiency virus infection (HIV)

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T. Teachey, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Teachey DT, Obzut DA, Axsom K, Choi JK, Goldsmith KC, Hall J, Hulitt J, Manno CS, Maris JM, Rhodin N, Sullivan KE, Brown VI, Grupp SA. Rapamycin improves lymphoproliferative disease in murine autoimmune lymphoproliferative syndrome (ALPS). Blood. 2006 Sep 15;108(6):1965-71. doi: 10.1182/blood-2006-01-010124. Epub 2006 Jun 6. PMID 16757690
- [Background] Teachey DT, Manno CS, Axsom KM, Andrews T, Choi JK, Greenbaum BH, McMann JM, Sullivan KE, Travis SF, Grupp SA. Unmasking Evans syndrome: T-cell phenotype and apoptotic response reveal autoimmune lymphoproliferative syndrome (ALPS). Blood. 2005 Mar 15;105(6):2443-8. doi: 10.1182/blood-2004-09-3542. Epub 2004 Nov 12. PMID 15542578
- [Result] Teachey DT, Greiner R, Seif A, Attiyeh E, Bleesing J, Choi J, Manno C, Rappaport E, Schwabe D, Sheen C, Sullivan KE, Zhuang H, Wechsler DS, Grupp SA. Treatment with sirolimus results in complete responses in patients with autoimmune lymphoproliferative syndrome. Br J Haematol. 2009 Apr;145(1):101-6. doi: 10.1111/j.1365-2141.2009.07595.x. Epub 2009 Feb 4. PMID 19208097
- [Result] Bride KL, Vincent T, Smith-Whitley K, Lambert MP, Bleesing JJ, Seif AE, Manno CS, Casper J, Grupp SA, Teachey DT. Sirolimus is effective in relapsed/refractory autoimmune cytopenias: results of a prospective multi-institutional trial. Blood. 2016 Jan 7;127(1):17-28. doi: 10.1182/blood-2015-07-657981. Epub 2015 Oct 26. PMID 26504182

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus Treatment
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11 [1.8 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 and 4 Toxicities of Administration of Oral Sirolimus
Description: Grade 3 toxicities are those that are considered severe or medically equivalent requiring hospitalization or prolonged hospitalization (according to CTCAE criteria 3.0).
  Grade 4 toxicities are those that are life-threatening (urgent intervention indicated) (according to CTCAE criteria 3.0).
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 30
participants | 1

2. Secondary Outcome: Number of Participants With Autoimmune Disease Response to Oral Sirolimus
Description: Complete response (CR) is complete resolution in all autoimmune cytopenias (neutropenia, anemia thrombocytopenia) maintained for more than two months, combined with an ability to wean off corticosteroids and/or other immunosuppressive medication. Partial response (PR) is improvement in any cytopenias by at least one grade, lasting more than two months, without worsening any other cytopenias or stable disease with the ability to wean corticosteroids and/or immunosuppressive medications by at least 50%. No response (NR) is no change in cytopenias with treatment, and the inability to wean corticosteroids or other immunosuppressive medications. Progressive disease (PD) refers to obtaining a CR or PR by the 3 month observation and relapsing or progressing by the 6 month observation, leading to cessation of study drug.
Time Frame: 6 months
Population: Number analyzed per row reflects number of participants with each condition
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 30
Participants
  Response in patients w/ ALPS: number analyzed (Participants) | 12
  Response in patients w/ ALPS: Complete Response (CR) | 11
  Response in patients w/ ALPS: Partial Response (PR) | 1
  Response in patients w/ ALPS: No Response (NR) | 0
  Response in patients w/ ALPS: Progressive Disease (PD) | 0
  Response in patients w/ multilineage cytopenias: number analyzed (Participants) | 12
  Response in patients w/ multilineage cytopenias: Complete Response (CR) | 7
  Response in patients w/ multilineage cytopenias: Partial Response (PR) | 1
  Response in patients w/ multilineage cytopenias: No Response (NR) | 2
  Response in patients w/ multilineage cytopenias: Progressive Disease (PD) | 2
  Resp pts w/ single-lineage autoimmune cytopenias: number analyzed (Participants) | 6
  Resp pts w/ single-lineage autoimmune cytopenias: Complete Response (CR) | 1
  Resp pts w/ single-lineage autoimmune cytopenias: Partial Response (PR) | 2
  Resp pts w/ single-lineage autoimmune cytopenias: No Response (NR) | 3
  Resp pts w/ single-lineage autoimmune cytopenias: Progressive Disease (PD) | 0

3. Secondary Outcome: Trough Levels Produced by Administration of Oral Sirolimus
Description: Pharmacokinetic levels produced by administration of oral sirolimus
Time Frame: Within first 5 days of starting sirolimus
Measure: Mean (Full Range); unit: nanograms/dL
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 30
nanograms/dL | 8.5 [2.9 to 20]

4. Secondary Outcome: Effect of Sirolimus on Intracellular Targets
Description: Needs more specific information
Time Frame: 6 months
Population: This was an optional assessment- there was no enrollment. Data were not collected.
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Lymphoproliferation Response to Oral Sirolimus
Description: Complete response (CR) is complete resolution of any lymphadenopathy and splenomegaly for at least two months. Partial response (PR) is a reduction in size of at least 50% of lymphadenopathy or splenomegaly for at least two months. No response (NR) is no change or < 50% reduction in lymphadenopathy or splenomegaly. Progressive Disease (PD) is obtaining a CR or PR by the 3 month observation and relapsing or progressing by the 6 month observation, leading to cessation of study drug. Not Applicable (N/A) is there is no evidence of disease (No pathologic lymphadenopathy or splenomegaly at time of enrollment).
Time Frame: 6 months
Population: Number analyzed per row reflects number of participants with each condition
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus Treatment
Number analyzed (Participants) | 30
Participants
  Response in patients w/ ALPS: number analyzed (Participants) | 12
  Response in patients w/ ALPS: Complete Response (CR) | 11
  Response in patients w/ ALPS: Partial Response (PR) | 1
  Response in patients w/ ALPS: No Response (NR) | 0
  Response in patients w/ ALPS: Progressive disease (PD) | 0
  Response in patients w/ ALPS: Not Applicable (N/A) | 0
  Response in patients w/ multilineage cytopenias: number analyzed (Participants) | 12
  Response in patients w/ multilineage cytopenias: Complete Response (CR) | 3
  Response in patients w/ multilineage cytopenias: Partial Response (PR) | 0
  Response in patients w/ multilineage cytopenias: No Response (NR) | 1
  Response in patients w/ multilineage cytopenias: Progressive disease (PD) | 1
  Response in patients w/ multilineage cytopenias: Not Applicable (N/A) | 7
  esp pts w/ single-lineage autoimmune cytopenias: number analyzed (Participants) | 6
  esp pts w/ single-lineage autoimmune cytopenias: Complete Response (CR) | 1
  esp pts w/ single-lineage autoimmune cytopenias: Partial Response (PR) | 0
  esp pts w/ single-lineage autoimmune cytopenias: No Response (NR) | 0
  esp pts w/ single-lineage autoimmune cytopenias: Progressive disease (PD) | 0
  esp pts w/ single-lineage autoimmune cytopenias: Not Applicable (N/A) | 5

ADVERSE EVENTS:
Arm/Group | Sirolimus Treatment
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 15/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Treatment (N=30)
Vasculitis (Nervous system disorders) | 1 (1) — This adverse event was determined not to be related to study treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Treatment (N=30)
Mucositis (Gastrointestinal disorders) | 10 (10)
Elevated triglycerides and cholesterol (Cardiac disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Sun sensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Gastro-esophageal reflux disease (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes